CLINICAL TRIAL: NCT01793636
Title: An Open Label, Randomised Phase II Study, Comparing AZD2014 Versus Everolimus With Advanced Metastatic Renal Cancer and Progression on VEGF Targeted Therapy
Brief Title: A Study Comparing AZD2014 vs Everolimus in Patients With Metastatic Renal Cancer
Acronym: ZEBRA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inferior efficacy of study drug in renal indication.
Sponsor: Queen Mary University of London (Other)
Collaborators: AstraZeneca (Industry); Cancer Research UK (Other)
Responsible Party: Principal Investigator, Centre of Experimental Medicine, Chief Investigator, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 008424 QM; NCT01996722 (obsolete NCT alias)
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Metastatic Clear Cell Renal Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — vistusertib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD2014 (Experimental): AZD2014- tablets, starting dose 50mg BD everyday, until disease progression or untolerable toxicity
  Interventions: Drug: AZD2014
- Everolimus (Active Comparator): Everolimus- tablets, starting dose 10mg OD everyday until disease progression or untolerable toxicity
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: AZD2014 — AZD2014 vs Everolimus
  Other Names: Everolimus/Afinitor
  Arms: AZD2014
Drug: Everolimus — comparing PFS in patients treated with AZD2014 vs Everolimus
  Other Names: Afinitor
  Arms: Everolimus

SUMMARY:
When kidney cancer spreads beyond the kidney, it is known as metastatic kidney cancer. This is very difficult to treat and almost all patients will die of their disease within 2 years of the diagnosis.

Sunitinib and other related drugs (e.g. pazopanib) have become standard therapy for untreated patients with metastatic kidney cancer. They target a growth factor known as VEGF which is important in treating kidney cancer. Although the results with this drug are impressive, patients develop resistance to the drug and stop therapy. It is currently standard practice is to give everolimus when resistance to sunitinib occurs; this is associated with clear clinical benefit.

However the average time to cancer regrowth with everolimus is only 5 months. It is thought this might be because, everolimus only partially inhibits its target (TORC 1 and TORC 2). Therefore further improvement in treating patients is required. AZD2014 is a promising new drug which does inhibit both TORC 1 and TORC 2 and is therefore worthy of investigation in renal cancer as it theoretically could may have advantages over everolimus. Therefore study compares AZD2014 to everolimus in the setting where everolimus is used as standard of care. (e.g. in patients who have failed drug like sunitinib). The study is a randomised trial allowing us to quantify the benefit and potential for further development of AZD2014. Repeat Xrays (CT scans) will be used to assess if the new drug delays tumour growth. Patients will be closely followed up in clinic to ensure safety. A maximum of 122 patients will be recruited into this multi centre national trial. The primary goal of the study is to investigate if AZ2014 delays the time for cancer regrowth (time to progression) compared to everolimus.

DETAILED DESCRIPTION:
Renal cell cancer, also referred to as kidney cancer, is diagnosed in approximately 170,000 people worldwide annually, resulting in 82,000 deaths. Treatment for metastatic kidney cancer is difficult. Almost all of the patients die from their disease.

In 2006 a new drug called sunitinib, a tyrosine kinase inhibitor, transformed treatment options. It targets the development of new blood vessels within the cancer. Although the results with this drug are impressive, patients develop resistance a median after 11 months to the drug, relapse and die of renal cancer. It is currently standard practice to switch to everolimus when resistance to sunitinib occurs; this is associated with clear clinical benefit.

POTENTIAL RISKS FOR PATIENTS RECEIVING AZD2014:

The main risks and burdens to the patients participating in the study are the potential for side effects of the AZD2014 drug. The phase I study using this drug has been completed, therefore we know it is safe to administer to patients and we have a good idea of what side effects the drug causes. But as the drug is given to larger numbers, additional side effects may be discovered. The activity of the drug has not been evaluated in kidney cancer. Therefore we are not sure if AZD2014 will work

POTENTIAL RISKS FOR PATIENTS RECEIVING EVEROLIMUS:

Everolimus is the current standard therapy for these patients so the risks associated with study drug for these patients are the same as standard of care.

POTENTIAL RISKS FOR ALL PATIENTS:

SIDE EFFECTS:

Side effects will be closely monitored during and after the study. Patients are required to attend clinic weekly for the first four weeks and then every 4 weeks whilst they are on study medication where adverse events will be recorded.

The patient information sheet includes details on expected adverse events for patients to look out for and also details that unexpected events may occur. Patients are provided with the research nurse and principal investigator contact details should any adverse events occur during the course of the study.

Other medical professionals are informed that patients are receiving an experimental drug (through GP letter and labelling of hospital records). There will be an independent data monitoring committee for the trial which will closely assess the side effects of the drugs on a regular basis and the trial results to make sure there are no risk excess to patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed renal cell carcinoma with measurable metastases on CT/MRI imaging. Only a component of clear cell is required.
2. Radiological progressive disease on VEGF targeted therapy (RECIST v1.1). Exposure to more than one line of VEGF targeted therapy is acceptable. Previous treatment with initial interferon or IL-2 or other experimental agent is acceptable (with the exception of drugs specifically targeting mTOR).
3. Evidence of measurable disease (ie, ≥1 malignant tumour mass that can be accurately measured in at least 1 dimension ≥ 20 mm with conventional computerized tomography [CT] scan or Magnetic Resonance Imaging [MRI], or ≥10 mm (except lymph nodes which must have short axis ≥ 15 mm) with spiral CT scan using a 5 mm or smaller contiguous reconstruction algorithm). Bone lesions, ascites, peritoneal carcinomatosis or miliary lesions, pleural or pericardial effusions, lymphangitis of the skin or lung, cystic lesions, or irradiated lesions are not considered measurable.
4. Adequate organ function as defined by the following criteria:

   1. Total serum bilirubin ≤1.5 x ULN (patients with Gilbert's disease exempt),
   2. Serum transaminases ≤3.0 x ULN (x5 in the presence of liver metastasis).
   3. Serum creatinine ≤ 2 x ULN or Cockcroft and Gault >30ml/min
   4. Absolute neutrophil count (ANC) ≥1.5 x 109/L without growth factor support,
   5. Platelets ≥ 100 x 109/L
5. Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrolment.
6. Willingness and ability to comply with scheduled visits, treatment plans and laboratory tests and other study procedures
7. ECOG performance status of 0, 1 or 2.
8. Life expectance >12 weeks
9. At least 14 days since the end of prior systemic treatment (sunitinib, pazopanib, sorafenib), radiotherapy, or surgical procedure with resolution of all treatment-related toxicity to NCI CTCAE Version 4.0 grade ≤1 or back to baseline except for alopecia or hypothyroidism. A 21 day gap between bevacizumab and interferon therapy should exist.
10. Fasting blood sugar ≤8mmol/l and HbA1C ≤7%
11. Age ≥18 years

Exclusion Criteria:

1. Previous exposure to mTOR inhibitors for metastatic renal cancer.
2. Females of child-bearing potential. The definition of child-bearing potential: women between menarche and menopause who have not been permanently or surgically sterilised and capable of procreation. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. Male patients must be surgically sterile or agree to use effective contraception.
3. Pregnant and Breast feeding women.
4. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormally that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgement of the investigator, would make the patient inappropriate for entry into this study. Specifically the following indications are contraindicated: Hereditary galacto-intolerance, glucose/galactose malabsorption and lactose deficiency
5. Untreated clinically symptomatic brain or meningeal metastases. Patients with evidence of clinically stable brain metastases are eligible providing that they do not require corticosteroids.
6. Any evidence of severe or uncontrolled diseases e.g., unstable or uncompensated respiratory, hepatic or renal disease.
7. Evidence of interstitial fibrotic lung disease (bilateral, diffuse, parenchymal lung disease).
8. Unresolved toxicity ≥ CTCAE v.4.0 grade 2 (except alopecia and hypothyroidism) from previous anti-cancer therapy.
9. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ or localised controlled prostate cancer) within 5 years, unless the patient has been disease free for 2 years and there is a tissue diagnosis of the primary cancer of interest from a target lesion.
10. Uncontrolled diabetes mellitus or hyperlipidaemia (> grade 1)
11. Treatment with an investigational drug (not including VEGF TKIs such as pazopanib/ tivozanib) within 21 days prior to the first dose of therapy. If investigational drug is a VEGF TKI then with 14 days prior to the first dose of therapy
12. Patients who have experienced any of the following procedures or conditions currently or in the preceding 12 months:

    1. Coronary artery bypass graft
    2. Angioplasty
    3. Vascular stent
    4. Myocardial infarction
    5. Angina pectoris
    6. Congestive heart failure new york heart association grade ≥2
    7. Ventricular arrhythmias requiring continuous therapy
    8. Supraventricular arrhythmias including atrial fibrillation, which are uncontrolled
    9. Haemorrhagic or thrombotic stroke, including transient ischaemic attacks or
    10. Any other central nervous system bleeding
13. Mean resting QTcF ≥470 msec as per local reading
14. Abnormal ECHO at baseline (left ventricular ejection fraction [LVEF] <50%
15. Known inherited or acquired immunodeficiency
16. Known active hepatitis B or C infection or Known HIV.
17. Other concomitant anti-cancer therapy (including LHRH agonists) except steroids
18. Previous bone marrow transplant
19. Age <18 years
20. Any haemopoietic growth factors (eg, G-CSF, GM-CSF) within 2 weeks prior to receiving study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
To investigate if single agent AZD2014 delays progression free survival compared to everolimus using RESIST v1.1 | Completion of study- approx 3 years

SECONDARY OUTCOMES:
To evaluate tumour response rate after at least 8 weeks of treatment with the study drugs. | 3 years

OTHER OUTCOMES:
To compare overall survival of the two group of patients. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Powles, Principal Investigator — Queen Mary University of London, UK
Locations (9):
- United Kingdom (9):
  - Royal Bournemouth Hospital, Bournemouth
  - Royal Sussex County Hospital, Brighton
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - Beatson West of Scotland Cancer Center, Glasgow
  - St. James' Hospital, Leeds
  - Barts Health NHS Trust, London
  - Royal Free London Hospital, London
  - Southampton General Hospital, Southampton
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea

REFERENCES:
- See also: Related Info — http://www.cancerresearchuk.org/cancer-help/